CLINICAL TRIAL: NCT03201991
Title: ALS Study Determining Various Biomarkers and Strength Comparison After Exercise
Acronym: ADVANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003843
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Program (Other): Participants will be asked to take part in an exercise program that is focused on quadriceps strengthening.
  Interventions: Other: Resistance Exercise Program

INTERVENTIONS:
Other: Resistance Exercise Program — The resistance exercise program will involve three sets of 10 repetitions of each exercise in levels 1 and 2 every day. Participants will be given instructions to follow.

SUMMARY:
The purpose of this study is to determine the muscle strength of a muscle in the thigh after 12 weeks of home exercise.

DETAILED DESCRIPTION:
Study participation lasts a total of three months and includes two study visits. Subjects are asked to undergo strength testing, physical exams, lab draws, and muscle biopsies at each study visit. Muscle biopsies are done in the quadriceps muscle. In between study visits, subjects are asked to maintain a weekly exercise regimen given to them by the study physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable or definite amyotrophic lateral sclerosis (ALS) based on the revised El-Escorial criteria
* Presence in ipsilateral leg of either weakness in any muscle group or of active denervation by needle electromyography (EMG) which is a surrogate marker of early denervation
* Ipsilateral quadriceps femoris strength: >=4
* Ambulatory with or without assistance
* Revised ALS Functional Rating Scale (ALSFRS-R) Score > 30
* Forced expiratory vital capacity (FVC) >50% of predicted

Exclusion Criteria:

* ALSFRS-R ≤ 30
* Quadriceps femoris strength <4
* Unable to walk or uses wheelchair as primary means of mobility
* More than mild atrophy of quadriceps
* Bleeding disorder or uptake of anticoagulants
* Unwilling to comply with exercise and needle muscle biopsy
* Not a good research candidate according to the medical opinion of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Change in functional muscle strength | Week 12
  determine the functional muscle strength of quadriceps femoris muscles before and after 12 weeks of home exercise

CONTACTS AND LOCATIONS:
Overall Officials: Omar Jawdat, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States